CLINICAL TRIAL: NCT03603730
Title: Modulation of Gastric Sensitivity and Accommodation by Vagal Nerve Stimulation
Brief Title: Vagal Nerve Stimulation for Functional Dyspepsia and Gastroparesis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Braden Kuo, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2010P000440
Record Dates: First submitted 2018-07-04; First posted 2018-07-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-05

CONDITIONS: Dyspepsia; Gastroparesis
Keywords: Functional Dyspepsia; Gastroparesis
MeSH Terms: conditions — Dyspepsia; Gastroparesis

STUDY DESIGN:
Intervention Model Description: There will be multiple study visits consisting of a screening, baseline testing, consumption of a liquid meal, and fMRI brain and gut imaging sessions. Visits will include active and inactive taVNS delivered to the outer ear at a moderate, non-painful level.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- taVNS (Experimental): Active or inactive taVNS
  Interventions: Device: taVNS

INTERVENTIONS:
Device: taVNS — Active or inactive taVNS delivered to the external ear at a moderate, non-painful level.

SUMMARY:
Explore the effects of auricular transcutaneous vagal nerve stimulation (taVNS) on brain and stomach outcomes in functional dyspepsia and gastroparesis patients.

DETAILED DESCRIPTION:
The primary aims of this study are to 1) investigate the effects of auricular transcutaneous vagal nerve stimulation (taVNS) on brain-gut signaling using a liquid meal test in functional dyspepsia (FD) and gastroparesis (GP) patients using combined gastric, autonomic and neuroimaging measures, and 2) evaluate the effectiveness of taVNS on FD and GP symptoms.

A total of 25 FD and 25 GP patients will be enrolled in this study, both females and males, ranging between 18 and 65 years of age. There will be multiple study visits consisting of a screening, baseline testing, consumption of a liquid meal, and fMRI brain and gut imaging sessions. Visits will include active and inactive taVNS delivered to the outer ear at a moderate, non-painful level.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers, female and male, between 18 and 65 years of age.
2. For healthy volunteers, ability to undergo MRI for up to 2 hours.
3. For Functional Dyspeptic patients, diagnosis according to the Rome III criteria for both PDS and EPS subtypes.
4. For Gastroparesis patients, diagnosis will include the following criteria:

   * symptoms of gastroparesis of at least 12 weeks duration (does not have to be continuous) with varying degrees of nausea, vomiting, early satiety, and/or post-prandial fullness
   * an idiopathic etiology
   * abnormal gastric emptying scintigraphy (GES) results using a 4 hour low fat Egg Beaters® protocol within the last 6 months with either a gastric emptying rate > 60% retention at 2 hours and/or >10% retention at 4 hours.

4) Stable medical treatment for Functional Dyspeptic or Gastroparesis during 1 month before study and during the study period.

5) Avoidance of alcohol, nicotine, and caffeine for 24 hours prior to study session.

Exclusion Criteria:

1. History gastric/esophageal surgery
2. Any alternative treatment (e.g. acupuncture, hypnosis etc.) two weeks prior to the study or during the study period.
3. Illicit drugs or opioid use.
4. History of arrhythmias.
5. Implanted pacemaker.
6. Epilepsy or a prior history of seizures.
7. For Gastroparesis patients, inability to comply with or complete GES test (including allergy to eggs).
8. Pregnancy or nursing or plans to become pregnant.
9. Inability to provide informed consent.
10. BMI more than 32 and/or weight > 235 lbs. (limits of the MRI table).
11. Contraindications for MRI: High magnetic fields may pose a serious health hazard to subjects with implanted ferromagnetic objects. Every subject in this study will be carefully screened before entering the high magnetic field shielded room to collect a precise outline of the subject's medical history. Subjects with the following characteristics/disease may not be eligible to participate in the study and will require additional screening:

    * History of Head Trauma
    * Any metallic implants (e.g. braces or permanent retainers)
    * Tattoos with metallic ink above the nipple line
    * Surgical Aneurysm Clips
    * Cardiac Pacemaker
    * Prosthetic Heart Valve
    * Neurostimulator
    * Implanted pumps
    * Cochlear Implants
    * Metal rods, Plates, Screws
    * Recent Previous Surgery
    * IUD
    * Hearing Aid
    * Dentures (which might create NMR artifacts)
    * Metal Injury to eyes
    * Pregnancy or plans to become pregnant
    * Breast Feeding
    * Meniere's Disease
    * Transdermal (skin) patches such as NicoDerm (nicotine for tobacco dependence), Transderm Scop, or Ortho Evra (birth control)
    * Claustrophobia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-11-30 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Neuroimaging | 2 hours
  Functional magnetic resonance imaging (fMRI)

SECONDARY OUTCOMES:
Electrogastrography (EGG) | 2 hours
  We will use EGG to measure slow wave myoelectrical activity, as measured by EGG power/peak frequency.
Electrocardiography (ECG) | 2 hours
  We will use ECG to examine high frequency heart rate variability (HF-HRV), i.e. the R-peak of the QRS complex.
Respiration | 2 hours
  Respiration will be measured in beats per minute (bpm).
Skin Conductance Levels (SCL) | 2 hours
  SCL will measured in volts per second.

OTHER OUTCOMES:
Liquid meal challenge | 40 minutes
  Patients will be studied in the morning after overnight fast. The liquid meal test will be conducted in the following way: subjects consume 120 ml of Ensure every 4 min until full. At 5 min intervals, participants score fullness using a rating scale that combines verbal descriptors on a scale graded 0-5. Participants are told to stop when a score of 5 is obtained.
Short Form Nepean Dyspepsia Index (SF-NDI) | 5 minutes
  Subjects will be asked to complete multiple questionnaires during the sessions, including the SF-NDI. The SF-NDI consists of 10 questions regarding the effects of dyspepsia symptoms ("stomach problems") on different aspects of life (tension, interference with daily activities, eating/drinking, knowledge/control, and work/study) as they pertain to the last week. Each response can be from 1 (not at all affected) to 5 (extremely affected), or 0 (N/A), for a total summed score out of 50.
Brief Pain Inventory (BPI) | 5 minutes
  Subjects will be asked to complete multiple questionnaires during the sessions, including the BPI. The BPI assesses the severity of the subject's pain as well as the degree of disability and impact on daily functioning over the past 24 hours and past 7 days. This questionnaire includes a diagram of the human body in which the subject would shade in where they feel pain, placing an X on the area that hurts the most, as well as series of questions rating the subject's pain from 0 (no pain) to 10 (pain as bad as you can imagine) and on the relief felt from treatments or medications as measured from 0% (no relief) to 100% (complete relief).
Visual Analog Scale (VAS) | 5 minutes
  Subjects will be asked to complete multiple questionnaires during the sessions, including the VAS. The VAS measures satiation, abdominal pain/discomfort, nausea, bloating, and belching on a visual scale (0-100mm) with the descriptors "unnoticeable" and "unbearable" as anchors for 0mm and 100mm respectively. It will be administered at multiple time points across a session, with the sum of the 0-100mm scales for each symptom providing an aggregate symptom score.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Sclocco, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No